CLINICAL TRIAL: NCT00520624
Title: Treatment of Exercise-induced Laryngo Obstruction in Elite Athletes
Brief Title: Treatment of Exercise-induced Laryngomalacia in Elite Athletes
Acronym: EIL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients willing to join
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Backer, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC-EIL-07-ELITE
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Exercise-induced Laryngomalacia
Keywords: EIL
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Treatment 1, for those with high degree of EIL
  Interventions: Device: inspiratory muscle strength training
- 2 (Experimental): Treatment 2, for those with high degree of EIL
  Interventions: Procedure: Surgery
- 3 (No Intervention): Control group of those with high degree of EIL
- 4 (Experimental): Treatment 1, for those with low degree of EIL
  Interventions: Device: inspiratory muscle strength training
- 5 (No Intervention): Control group of those with low degree of EIL

INTERVENTIONS:
Device: inspiratory muscle strength training
  Arms: 1; 4
Procedure: Surgery
  Arms: 2

SUMMARY:
Treatment of exercise-induced laryngomalacia (an obstruction of larynx during physical activity) in elite athletes using two different treatments. The study is randomized with control groups.

ELIGIBILITY:
Inclusion Criteria:

* Laryngoscopically verified EIL,
* Elite athlete for a minimum of 1 year and continuing for a minimum 6 months after start of treatment

Exclusion Criteria:

* Has to be able to run on treadmill

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Lungemedicinsk Forskningsenhed, Copenhagen, Denmark